CLINICAL TRIAL: NCT06206876
Title: First-in-Human Phase I Trial of FL118 in Patients With Advanced Pancreatic Ductal Adenocarcinoma
Brief Title: FL118 for Treating Patients With Advanced Pancreatic Ductal Adenocarcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: never opened
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I 3555023; NCI-2023-08681 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 3555023 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2023-12-06; First posted 2024-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Advanced Pancreatic Ductal Adenocarcinoma; Locally Advanced Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Refractory Pancreatic Ductal Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; Specimen Handling; 7-ethyl-7-hydroxy-10H-1,3-Dioxolo(4,5-g)pyrano(3',4':6,7)indolizino(1,2-b)quinoline-8,11(7H,12H)-dione; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (FL118) (Experimental): Patients receive FL118 PO on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and CT or MRI throughout the trial. Patients may optionally undergo biopsy at screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: DDX5 Degrader FL118; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: DDX5 Degrader FL118 — Given PO
  Other Names: FL 118; FL-118; FL118
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of FL118 in treating patients with pancreatic ductal adenocarcinoma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). FL118 is a small anti-tumor molecule that inhibits the expression of multiple cancer-associated anti-apoptotic proteins. An anti-apoptotic protein is a protein that interferes with or inhibits cell death. In adults, apoptosis is used to rid the body of cells that have been damaged beyond repair. Apoptosis also plays a role in preventing cancer. If apoptosis is for some reason prevented, it can lead to uncontrolled cell production that can subsequently develop into a tumor. FL118 has been shown to inhibit or block the proteins that prevent damaged/mutated (genetically changed) cells from dying, and, by doing so, prevent the growth of cancerous cells and tumor development.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety, schedule, and dosing of DDX5 degrader FL118 (FL118) in patients with advanced pancreatic ductal adenocarcinoma (PDAC).

II. To determine the pharmacokinetics (PK) of FL118 in patients with advanced PDAC.

SECONDARY OBJECTIVES:

I. To determine the pharmacodynamics (PD) of FL118 in patients with advanced PDAC.

II. To determine the preliminary antineoplastic efficacy of FL118 in patients with advanced PDAC.

EXPLORATORY OBJECTIVES:

I. To evaluate biomarkers predictive of response or resistance. II. Evaluate changes in the tumor microenvironment. III. To determine the significance of somatic and germline DNA damage repair mutations as predictive biomarkers of antineoplastic activity.

OUTLINE: This is a dose-escalation study of FL118 followed by a dose-expansion study.

Patients receive FL118 orally (PO) on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial. Patients may optionally undergo biopsy at screening and on study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Have a histologically or cytologically confirmed advanced PDAC (locally advanced/unresectable or metastatic for part A (dose escalation) and metastatic for part B (dose expansion)
* Progression on or intolerance to 1st line therapy for advanced disease. Note that completion of adjuvant or neoadjuvant chemotherapy within 6 months from relapsed disease is considered one line of therapy for locally advanced/unresectable or metastatic disease
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have a life expectancy of greater than 3 months
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Patient willing to undergo tumor biopsy at baseline and on treatment if there is a lesion that can safely be biopsied based on investigator assessment. If this is not feasible, adequate archival tumor tissue must be available
* Absolute neutrophil count (ANC): ≥ 1,500/mL
* Platelets: ≥ 100,000/mL
* Hemoglobin: ≥ 9 g/dL
* Creatinine clearance ≥ 60 mL/min (per Cockroft-Gault equation)
* Total bilirubin: ≤ 1.5 X upper limit of normal (ULN) or, direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): ≤ 2.5 X ULN or, ≤ 5 X ULN for subjects with liver metastases
* Albumin: ≥ 3 gm/dL
* For females of reproductive potential (those who have not been surgically sterilized or have not been free from menses for > 1 year): use of highly effective contraception for at least 1 month prior to screening and agree to use such a method during study participation and, for an additional 6 months after the end of FL118 oral administration
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during the study participation and for an additional 3 months after the end of FL118 oral administration
* Be willing and able to comply with all study procedures and, availability for the duration of the study
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Has a major surgical procedure within 4 weeks prior to the planned first day of study drug dosing
* Received a prior treatment intended for antitumor effect (medication, surgery, radiotherapy, etc.) within 2 weeks prior to the planned first day of study drug dosing (or patient who received mitomycin C or nitrosourea within 6 weeks prior to the planned first day of study drug dosing)
* Has an active infection requiring systemic therapy
* Has a history of organ transplantation
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through the trial period after the last dose of trial treatment
* Has congestive heart failure (class III or IV New York Heart Association), acute coronary syndrome, acute cerebrovascular episode, acute peripheral vascular disease, or clinically significant cardiac arrhythmia within 6 months prior to the planned first day of study drug dosing
* Has clinically significant venous thromboembolic event (VTE), defined as lower extremity deep venous thrombosis or pulmonary embolism, within the past 3 months. Patients who are on a stable anticoagulant dose for VTE prophylaxis or treatment for at least 14 days are allowed to participate
* Bowel obstruction or perforation within the past 3 months
* Refractory malignant ascites or pleural effusions (requiring weekly para- or thoracentesis or indwelling catheter for palliation). Patients with less frequent/as needed para- or thoracentesis are allowed to participate
* Has difficulty taking oral medications, a digestive malabsorptive condition other than pancreatic exocrine insufficiency controlled with pancreatic enzyme replacement, or concurrent disease that significantly affects gastrointestinal function
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  Toxicity and adverse events will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Maximum tolerated dose (MTD) | 4 weeks from administation
  The MTD will be determined from the observed dose limiting toxicities per cohort using an accelerated dose-escalation design.
Recommended phase 2 dose | 4 weeks from administration
  The recommended phase 2 dose will be determined based on the MTD (or highest dose administered if the MTD is not reached), the pharmacokinetic/pharmacodynamic modeling, and overall clinical safety and efficacy data.
Half life | On days 1, 2, 15, and 16 of cycle 1 in dose-escalation phase
  PK parameters of half-life area
Maximum plasma concentration | On days 1, 2, 15, and 16 of cycle 1 in dose-escalation phase
  PK parameters of maximum plasma concentration
Area under the curve | On days 1, 2, 15, and 16 of cycle 1 in dose-escalation phase
  PK parameter area under the curve
CL/F | On days 1, 2, 15, and 16 of cycle 1 in dose-escalation phase
  apparent clearance of the analyte in the plasma

SECONDARY OUTCOMES:
Pharmacodynamics parameters | At baseline and cycle 2 day 23
  Will be collected at baseline and day 23
Overall response rate | Up to 12 months
  Will be assessed use a two-stage, single-arm Simon minimax design.
Disease control rate | Up to 12 months
  The disease control (complete response + partial response + stable disease) will be summarized using frequencies and relative frequencies. The disease control rate will be estimated with a 95% credible region obtained by Jeffrey's prior method.
Progression-free survival | From treatment until disease progression, death from disease, or last follow up, assessed up to 12 months
  Will be summarized using standard Kaplan-Meier methods, where estimates of median survival will be obtained with 95% confidence intervals.
Overall survival | From treatment until death due to any cause or last follow up, assessed up to 12 months
  Will be summarized using standard Kaplan-Meier methods, where estimates of median survival will be obtained with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States